CLINICAL TRIAL: NCT04492371
Title: COVID-19 INFECTION IN MULTIPLE MYELOMA PATIENTS: AN EUROPEAN OBSERVATIONAL STUDY
Brief Title: COVID-19 Infection and Multiple Myeloma
Acronym: EMN-COVID
Status: Completed | Type: Observational
Sponsor: Stichting European Myeloma Network (Network)
Collaborators: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Organization: European Myeloma Network B.V. (Network)
Other Study IDs: EMN-COVID
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma; Covid19; Corona Virus Infection
MeSH Terms: conditions — Multiple Myeloma; COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Collect in an observational study the outcomes of COVID19 infection in MM patients across Europe.

DETAILED DESCRIPTION:
Coronavirus Disease 2019 (COVID-19), caused by a novel coronavirus (SARS-CoV-2), is a highly contagious disease that appeared in Wuhan, Hubei province of China in December 2019. It has now spread to multiple countries through infected persons travelling mainly by air. Most of the infected patients have mild symptoms including fever, fatigue and cough. But in severe cases, patients can progress rapidly and develop the acute respiratory distress syndrome, septic shock, metabolic acidosis and coagulopathy including a disseminated intravascular coagulation (DIC).

Multiple myeloma (MM) is a mature B-cell malignancy largely affecting the older patient with a median age at presentation of 70 years. The general performance status (PS) and the presence of comorbidity can identify a group of patients with poor tolerance to treatment, as well as risks of both bacterial and viral infection. MM patients have benefited significantly from therapeutic developments, however, the host response biology of the older person, coupled with a distinct disease biology overlay induces immune dysfunction. For example, the impact of aging on the human immune system is well documented. In MM it has long-since been understood that there is a spectrum of immune dysregulation, an important host factor considered in the "Hallmarks of cancer" theory. In addition, the delivery of anti-MM therapy includes immune modulating agents such as steroids, proteasome inhibitors and CD38-directed therapy though not all immune modulation is necessarily detrimental.

As such, myeloma patients are considered a higher risk in the current pandemic with SARS-COVID19. However, it is not clear whether this is actually the case, and the risk may not be different to population in general. Equally it may be sub-groups of patients who are at risk e.g. on treatment versus stable response (plateau), frailty. AS such, this proposal aims to collect in an observational study, the outcomes of COVID19 infection in MM patients across Europe.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Myeloma patients
* COVID-19 infection

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Multiple Myeloma patients with COVID-19 infection
Sampling Method: Probability Sample
Enrollment: 1054 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Nature of COVID19 | 1 years
  The duration of infection.
Costs related to COVID-19 | 1 years
  Costs related to Covid in terms of health resource needs.
Systemic anti-cancer therapy subgroup | 1 years
  Number of infection recovery for each systemic anti-cancer subgroup.
Laboratory values collected at hospitalization | 1 years
  Evaluate if recurring haematological and chemistry values are related to infection onset, better or poorer outcome.
COVID-19 infection in myeloma patient subgroups | 1 years
  Number of infection in each myeloma patient subgroups and evaluation of the number of recovery per subgroup.
Incidence of COVID-19 infection in frail patients | 1 years
  Number of frail patients with COVID-19 infection and resolution of it.
Infection outcome in different countries | 1 years
  Number of infection and outcome per country.

CONTACTS AND LOCATIONS:
Locations (8):
- General Hopspital Vienna/Medical University, Vienna, Austria
- UCL Saint-Luc, Brussels, Belgium
- University Hospital Ostrava, Ostrava, Czechia
- University Hospital Würzburg, Würzburg, Germany
- Alexandra Clinical Terapeutics, Athens, Greece
- AOU Consorziale Policlinico di Bari, Bari, Italy
- Amsterdam UMC, Amsterdam, Netherlands
- St James's University Hospital, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided